CLINICAL TRIAL: NCT07196735
Title: Bio-electrical Impedance Analysis in Patients With Functional Dyspepsia
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: BIA in FD
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Functional Dyspepsia; BIA; Fat Free Mass; Fat Mass; Phase Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with FD
- healthy patients

SUMMARY:
The primary objective of this study is to compare the BIA parameters, including Phase Angle, Fat Free Mass and Fat Mass, between women with functional dyspepsia and healthy women. All woman will undergo a bio-electrical impedance monitoring for this.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 - 75 years
* Fulfilling the ROME IV criteria for functional dyspepsia (for FD patients)
* FD unexplained by upper GI endoscopy during the past 12 months (mild gastritis allowed) (for FD patients).

Exclusion Criteria:

* Clinical suspicion of an organic disorder different from FD (patients can be included when this disorder had been excluded);
* Abnormality on upper GI endoscopy other than mild gastritis (for FD patients).
* Known reflux oesophagitis Los Angeles grade C or D, known Barrett oesophagus, peptic stricture.
* H pylori infection, unless treated at least 6 months before;
* Known inflammatory bowel disorder;
* Known major intestinal motility disorder;
* Alcohol (defined as more than 14 U per week) or other substance abuse;
* Active psychiatric disorder;
* Known systemic or auto-immune disorder with implication for the GI system;
* Prior abdominal surgery (with the exception of cholecystectomy or ap-pendectomy);
* Any prior diagnosis of cancer other than basocellular carcinoma;
* Current chemotherapy;
* History of gastro-enteritis in the past 12 weeks;
* Dietary supplements unless taken at a stable dose for more than 12 weeks;
* Treatment with neuromodulators (one neuromodulator taken at a sta-ble dose for more than 12 weeks is allowed);
* Treatment with PPI's during the past 8 weeks
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: female patients with or without FD between 18 and 75 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference in phase angle between healthy patients and patients with FD | from signing of the ICF till end of study (on average 1 week)
Difference in fat mass between healthy patients and patients with FD | from signing of the ICF till end of study (on average 1 week)
Difference in fat free mass between healthy patients and patients with FD | from signing of the ICF till end of study (on average 1 week)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No